CLINICAL TRIAL: NCT03359915
Title: Global Excellence in COPD Outcomes: Implementation and Effectiveness of COPD Self-Management Action Plans in Low and Middle Income Countries
Brief Title: GECo: Implementation and Effectiveness of COPD Self Management Action Plans in Low and Middle Income Countries
Acronym: GECo2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Collaborators: Johns Hopkins University (Other); Universidad Peruana Cayetano Heredia (Other); Asociacion Benefica Prisma (Other); Makerere University (Other); University of York (Other); Institute of Medicine, Tribhuvan University, Nepal (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16/0630_RCT
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Self-Management; Action Plan; SGRQ; LMIC; COPD Diagnosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: RCT Phase - Parallel Groups: 240 in total Control arm - 120 participants Intervention Arm - 120 participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patient education in use of a COPD self-management action plan supported by monthly visits from, and access to, a CHW who has been trained in the use of a COPD self-management action plan.
  Interventions: Behavioral: COPD Self-Management Plan
- Control Group (No Intervention): COPD 'standard' care in local setting - Bhaktapur, Nepal; Lima, Peru; Nakaseke, Uganda

INTERVENTIONS:
Behavioral: COPD Self-Management Plan — Patient education in use of a COPD self-management action plan supported by monthly visits from, and access to, a CHW who has been trained in the use of a COPD self-management action plan.
  Arms: Intervention Group

SUMMARY:
This study will randomise people with clinically significant COPD (GOLD Grade B-D) to usual care or provision of a self-management action plan supported by monthly follow-up visits from a community health worker trained in the use of the action plan. The primary outcome will be health-status: a comparison of the change in St. George's Respiratory Questionnaire (SGRQ) between baseline and 12 months in the two groups. We will randomise 240 people from three low- and middle-income countries, namely Nepal, Peru and Uganda. We will also examine the feasibility of implementing our self-management action plan intervention at scale.

DETAILED DESCRIPTION:
The investigators will determine whether a self-directed COPD Action Plan for the management of COPD exacerbations can be implemented with trained community health workers (CHWs). The investigators hypothesise that COPD action plans with disease-specific education and support from a CHW will lead to improved quality of life and will be locally-appropriate, acceptable, and feasible to implement.

1. Clinical Aim 1: Assess the clinical effectiveness of CHW-supported COPD Action Plans in LMICs by comparing change in disease-specific quality of life measures (SGRQ) at one year.
2. Implementation Aim 1: Assess the appropriateness, acceptability, and feasibility of implementing a CHW-supported, self-directed COPD Action Plan for management of COPD exacerbations.

The investigators will also determine whether a CHW-supported, self-directed COPD Action Plan is cost-effective, accounting for implementation realities. We hypothesise that COPD Action Plans are a cost-effective intervention, as measured by the incremental QALY.

1. Clinical Aim 2: Assess the cost-effectiveness of COPD Action Plans in terms of health-related costs and health benefits and explore broader cost implications to productivity.
2. Implementation Aim 2: Explore how the value of the COPD Action Plans is affected by both implementation factors that restrict optimal provision ('constraints') and sub-group differences, which have implications for equity.

The final design of our intervention will be informed by formative work prior to commencement of the main study.

Study fieldworkers will enroll and randomise 80 adults aged ≥40 years with GOLD GRADE B-D COPD at each of the following three countries in the catchment areas of existing community census areas in Bhaktapur (Nepal), Lima (Peru), and Nakaseke (Uganda). They will then be randomised via an online system into either a control (usual care) or intervention group.

The intervention arm will receive a specific self-management plan for COPD facilitated by trained CHWs, who will then visit the participants monthly. The control group will receive basic COPD education and be reminded about the sites for their local health care providers. The primary effectiveness outcome for the study will be change in health-status (SGRQ) between baseline and 12 months, across the two groups. We will also examine the cost-effectiveness of self-management for individuals with COPD.

The investigators will also examine the feasibility of implementing our self-management action plan intervention at scale.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥40 years
* Full-time resident in the area (living in area > 6 months)
* Able to perform adequate quality spirometry
* Capable of providing informed consent
* Identified as having COPD grade B-D as per GOLD criteria

Exclusion Criteria:

* Pregnancy (self-reported)
* Currently has active pulmonary TB or is taking medications for pulmonary TB
* Identified as having COPD grade A as per GOLD criteria

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Change in SGRQ | 12 months
  Comparison of the change in SGRQ between baseline and 12 months, in the intervention compared to the control arm.
  b) Implementation Aim 1: Assess the appropriateness, acceptability and feasibility of using questionnaires and PEF to identify COPD cases from the perspective of local community members, community health workers, local health centre physicians and ministries of health.

SECONDARY OUTCOMES:
Number of Exacerbations | 12 months
  Comparison of the number of COPD exacerbations in 12 months, between the intervention compared to the control arm.
Number of Hospitalisations | 12 months
  Comparison of the number of hospitalisations in 12 months, between the intervention compared to the control arm.
Number of CHW visits | 12 months
  Comparison of the number of CHW visits in 12 months, between the intervention compared to the control arm.
Health-Economics | 12 months
  Assess the cost-effectiveness of a supported COPD Action Plan in terms of health-related costs and health benefits and explore broader cost implications to productivity.

CONTACTS AND LOCATIONS:
Overall Officials: John R Hurst, FRCP, PhD, Principal Investigator — University College, London
Locations (3):
- Institute of Medicine, Kathmandu, Nepal
- Universidad Peruana Cayetano Heredia, Lima, Peru
- Makerere University Lung Institute, Makerere, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pollard SL, Siddharthan T, Hossen S, Rykiel NA, Flores-Flores O, Alupo P, Quaderi S, Ascencio I, Barber JA, Chandyo R, Das SK, Gianella G, Kirenga B, Grunstra K, Miranda JJ, Mohan S, Ricciardi F, Sharma AK, Shrestha L, Soares MO, Wosu AC, Hurst JR, Checkley W; GECo2 Trial Investigators. Chronic Obstructive Pulmonary Disease Self-Management in Three Low- and Middle-Income Countries: A Pilot Randomized Trial. Am J Respir Crit Care Med. 2023 Nov 15;208(10):1052-1062. doi: 10.1164/rccm.202303-0505OC. PMID 37698443
- [Derived] Siddharthan T, Pollard SL, Quaderi SA, Mirelman AJ, Cardenas MK, Kirenga B, Rykiel NA, Miranda JJ, Shrestha L, Chandyo RK, Cattamanchi A, Michie S, Barber J, Checkley W, Hurst JR; GECo Study Investigators. Effectiveness-implementation of COPD case finding and self-management action plans in low- and middle-income countries: global excellence in COPD outcomes (GECo) study protocol. Trials. 2018 Oct 19;19(1):571. doi: 10.1186/s13063-018-2909-8. PMID 30340648
- See also: The Johns Hopkins Center for Global NCD Research and Training Website — https://www.globalncd.org/
- See also: Trial Twitter account - @COPDGECo — https://twitter.com/copdgeco?lang=en